CLINICAL TRIAL: NCT03435302
Title: A Multicenter, Randomized, Controlled, Phase III Trial Comparing High-Dose IFN-a2b With Temozolomide Plus Cisplatin as Systemic Adjuvant Therapy for Resected Mucosal Melanoma
Brief Title: HDI Versus Chemotherapy as Systemic Adjuvant Therapy for Resected Mucosal Melanoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Lu Si, professor, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCHMMAT001
Record Dates: First submitted 2014-02-08; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Melanoma
Keywords: Mucosal Melanoma,Adjuvant Therapy,IFN-a2b,Temozolomide
MeSH Terms: conditions — Melanoma | interventions — Temozolomide; Cisplatin; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Temozolomide Plus Cisplatin (Experimental): per os 200 mg/m^2/d temozolomide on days 1 to 5 plus i.v. 75 mg/m^2 cisplatin divided into 3 days,which was repeated every 3 weeks for six cycles
  Interventions: Drug: Temozolomide Plus Cisplatin
- High-Dose IFN-a2b (Active Comparator): Participants will be treated with i.v. 15×10^6U/m^2/d IFN-a2b on days 1 to 5 each week for 4 weeks, followed by s.c. 9×10^6U IFN- a2b three times per week for 48 weeks.
  Interventions: Drug: High-Dose IFN-a2b

INTERVENTIONS:
Drug: Temozolomide Plus Cisplatin — Temozolomide is the oral analog of dacarbazine (DTIC), shows potential advantages over dacarbazine.
  Cisplatin is an agent that can potentially enhance the activity of temozolomide.
  Other Names: Temodal.; cisplatinum
  Arms: Temozolomide Plus Cisplatin
Drug: High-Dose IFN-a2b — Interferon belongs to the large class of glycoproteins known as cytokines.
  Other Names: Intron
  Arms: High-Dose IFN-a2b

SUMMARY:
This is a a multicenter, randomized, controlled, phase III trial comparing High-Dose IFN-a2b with Temozolomide Plus Cisplatin as Systemic Adjuvant Therapy for Resected Mucosal Melanoma.The study objective is to compare efficacy and safety of High-dose IFN-a2b and temozolomide-based chemotherapy as adjuvant therapy.

DETAILED DESCRIPTION:
The patients who comply with the inclusion and exclusion criteria will be enrolled. The estimated recruiting duration is 36 months. Patients with resected mucosal melanoma were randomized into two groups: HDI group (group A, treated with i.v. 15×10^6U/m^2/d IFN-a2b on days 1 to 5 each week for 4 weeks, followed by s.c. 9×10^6U IFN-a2b three times per week for 48 weeks), and chemotherapy group (group B, per os 200 mg/m^2/d temozolomide on days 1 to 5 plus i.v. 75 mg/m^2 cisplatin divided into 3 days,which was repeated every 3 weeks for six cycles). All patients will be followed for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than 18 years;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
3. Pathologically confirmed diagnosis of mucosal melanoma;
4. Completely resected primary tumor (once regional lymph nodes were involved, diagnosed by clinical or imaging examinations, lymphadenectomy was conducted);
5. No prior systemic adjuvant therapy or regional radiotherapy;
6. No evidence of distant metastatic disease evaluated by means of lymph nodes ultrasound, endoscopy, and ultrasound of anorectum and genitourinary tract, single-photon emission computed tomography (CT) of bone, and whole-body spiral CT or positron emission tomography-CT (PET-CT);
7. Normal bone marrow function; and adequate liver and renal function [including white blood cell (WBC) count > 3,000/mm^3;absolute neutrophil count > 1,500/mm^3; platelets >100,000/mm^3; serum creatinine less than two times of the upper limit of normal (ULN); bilirubin less than 1.5 times of ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 times of ULN; international normalized ratio less than 1.5 times of ULN; and partial thromboplastin time less than ULN].

Exclusion Criteria:

1. Cutaneous melanoma or ocular melanoma or melanoma of unknown primary site;
2. Incomplete resection or primary tumor unable to be resected;
3. A second cancer diagnosis;
4. Definite medical history of cirrhoses of the liver or autoimmune diseases;
5. Severe depression; and pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2014-02; Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) of high-dose IFN-a2b (HDI) and temozolomide-based chemotherapy as adjuvant therapy for resected mucosal melanoma. | Participants will be followed for an expected average of 24 months

SECONDARY OUTCOMES:
Distant metastasis-free survival(DMFS) of high-dose IFN-a2b (HDI) and temozolomide-based chemotherapy as adjuvant therapy for resected mucosal melanoma. | Participants will be followed for an expected average of 24 months
Overall survival (OS) of high-dose IFN-a2b (HDI) and temozolomide-based chemotherapy as adjuvant therapy for resected mucosal melanoma. | From date of randomization until the date of death from any cause, assessed up to 48 months
Number of Participants with Adverse Events of high-dose IFN-a2b (HDI) and temozolomide-based chemotherapy as adjuvant therapy for resected mucosal melanoma | Participants will be followed for the duration of hospital stay, an expected average of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China